CLINICAL TRIAL: NCT00187044
Title: Evaluation of the Safety of a Polyvalent Vaccinia Virus-HIV-1 Envelope Recombinant Vaccine (PolyEnv1) in Healthy Adults
Brief Title: Evaluation of the Safety of a Polyvalent Virus in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DID955; PolyEnv1; IND 7097
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2011-06

CONDITIONS: HIV Infection; Human Immunodeficiency Virus
Keywords: Vaccine; Prevention; HIV; AIDS
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Biological: PolyEnv1 vaccine

INTERVENTIONS:
Biological: PolyEnv1 vaccine — administered subcutaneously as 10*7 pfu in 0.8 mL

SUMMARY:
This is a research study to evaluate the safety of a vaccine to protect people from HIV infection. Human Immunodeficiency Virus (HIV) is the cause of AIDS (Acquired Immune Deficiency Syndrome). AIDS is one of the most serious viral infections of our time. It is believed that all persons who contract HIV will eventually develop AIDS. Because of this, we are trying to develop new ways to prevent infection with HIV.

The vaccine that will be tested in this study has been prepared from a small part of the HIV. The part of the HIV used in this vaccine is the "envelope" or coating part of the virus. In this study, researchers will evaluate how well the vaccine is tolerated, how much vaccine should be given, and determine if any side effects occur in response to the vaccination.

DETAILED DESCRIPTION:
This is a research study to evaluate the safety of a vaccine to protect people from HIV infection. Human Immunodeficiency Virus (HIV) is the cause of AIDS (Acquired Immune Deficiency Syndrome). AIDS is one of the most serious viral infections of our time. It is believed that all persons who contract HIV will eventually develop AIDS. Because of this, we are trying to develop new ways to prevent infection with HIV.

Vaccines have been very successful in preventing or decreasing the symptoms of a number of other viral infections such as hepatitis B, polio, and measles. Viral vaccines work by causing a person's immune system to make antibodies and immune cells against the virus or to "respond" to the virus. Because of the success with other viral infections, scientists are trying to develop a successful vaccine for HIV.

The vaccine that will be tested in this study has been prepared from a small part of the HIV. The part of the HIV used in this vaccine is the "envelope" or coating part of the virus. Because only this one part of the virus is used in the vaccine, the vaccine cannot cause HIV infection. The "envelope" part of HIV has been put into another virus, the vaccinia virus. The vaccinia virus has been used as a vaccine for many decades in millions of people and is the vaccine that eliminated the disease known as smallpox (i.e. smallpox vaccine). The smallpox vaccine is a licensed and effective vaccine. Making a new vaccine by putting part of a different virus into the smallpox vaccine (also known as vaccinia virus) is called a "recombinant" vaccinia virus vaccine. Our new recombinant vaccine product is called PolyEnv1. In this study, researchers will evaluate how well the vaccine is tolerated, how much vaccine should be given, and determine if any side effects occur in response to the vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults; age > 18 years, date of birth > 1972
* HIV-1 negative as documented by ELISA and Western blot analysis within 4 weeks immunization
* Normal history and physical exam
* Lower risk sexual behavior as defined by AVEG
* Normal complete blood count and differential defined as:
* hemoglobin > 11.0 gm/dl
* white blood cell count greater than or equal to 2500 cells/mm3
* platelet count between 150,000 and 550,000 cells/mm3
* total lymphocyte count greater than or equal to 650 cells/mm3
* CD4+ T cell count greater than or equal to 400 cells/mm3 Normal AST and ALT (<1.5 x the laboratory upper normal limit) and creatinine < 1.1 X ULN Normal CPK-MB (creatine kinase isoenzyme MB) and troponin I Normal ECG Negative PPD Availability for one year of follow-up No evidence of smallpox vaccination (born in the USA after 1972 with no detectable scar (on the deltoid, ankle, thigh or between the scapulae), and no history of vaccination in personal immunization record) No entry into military service before 1990 Informed consent

Fewer than 3 of the following:

Current cigarette smoker History of high cholesterol History of diabetes or high blood sugar High blood pressure Heart disease before age 50 in parent or sibling Vaccinia virus seronegative

Exclusion Criteria:

* History of immunosuppressive illness, chronic illness, or use immunosuppressive medications (e.g. steroids) or treatments
* Medical or psychiatric condition or occupational responsibilities which preclude subject compliance with the protocol. Specifically excluded are persons with a history of suicide attempts, recent suicidal ideation or who have past or present psychosis
* Subjects with identifiable higher risk behavior for HIV infection as determined by screening questions designed to identify risk factors for HIV infection. Specific exclusions include:
* History of injection drug use within the last 12 months prior to enrollment
* Higher or intermediate risk sexual behavior as defined by the AVEG
* Live attenuated vaccines within 60 days of study (subunit or killed vaccines [e.g. influenza or pneumococcal] are not exclusionary, but should be given at least 2 weeks away from HIV immunization)
* Use of experimental agents within 30 days prior to study
* Receipt of blood products or immunoglobulin in the past 6 months
* History of eczema, atopic dermatitis and other acute, chronic or exfoliative conditions
* Pregnant or lactating women
* Household contact with persons with immunodeficiency (including eczema or use of immunosuppressive medications)
* Household contact with persons less than 12 months of age
* Household contact with pregnant women
* Subjects with serious, life-threatening allergies to the antibiotic gentamicin
* Refusal of women to practice birth control for 3 months following vaccination.
* Known cardiac disease such as previous myocardial infarction, angina, congestive heart failure, or cardiomyopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 1997-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To determine the safety of PolyEnv1 administered via the subcutaneous route | 1 year

SECONDARY OUTCOMES:
To determine the maximum tolerated dose of PolyEnv1 and to evaluate the body's immune response to the vaccine | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pat Flynn, M.D., Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org